CLINICAL TRIAL: NCT00368121
Title: Phase II Study of Cetuximab for the Refractory or Relapsed Multiple Myeloma EMMA-1(Erbitux for Multiple Myeloma)
Brief Title: EMMA-1 (Erbitux for Multiple Myeloma)
Acronym: EMMA-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitable patients
Sponsor: Prof. Dr. Andreas Engert (Other)
Collaborators: The Clinical Trials Centre Cologne (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Andreas Engert, Prof. Dr., University of Cologne
Organization: University of Cologne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMMA-1
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cetuximab
MeSH Terms: conditions — Multiple Myeloma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab + Dexamethasone (Experimental)
  Interventions: Drug: Cetuximab +/- Dexamethasone

INTERVENTIONS:
Drug: Cetuximab +/- Dexamethasone — Cetuximab dosing schedule:
  • Loading dose of 400 mg/m2, followed by weekly doses of 250 mg/m2. Cetuximab will be administered once weekly over 16 weeks. Mode of administration: intravenous infusion
  Dexamethasone dosing schedule:
  • 20 mg administered on day 1-3, q1w, starting week 5 if evidence of tumor progression or week 9 if no PR or CR to Cetuximab alone.
  Mode of administration: orally
  Other Names: Erbitux

SUMMARY:
EMMA-1 is an open-label, non-randomized, two-stage phase II study. Patients with refractory multiple myeloma stage II or III or relapsed disease after at least one line of treatment will receive Cetuximab+/-Dexamethasone.

The planed treatment duration per patient is 16 weeks. Patients achieving a response or stable disease after 16 weeks of treatment may continue study medication for 6 more months (patients receiving Cetuximab alone) or for 3 more months (patients receiving Cetuximab plus Dexamethasone). Responding patients who relapse during follow-up period of two years may receive a second treatment with Cetuximab following initial study guidelines

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma diagnosed according to the Durie-criteria in stage II or III (Salmon and Durie)
* Measurable disease
* Refractory or relapsed disease after at least one line of treatment
* Male or female >= 18 years of age
* Life expectancy > 12 weeks
* ECOG performances status 0-2
* If of childbearing potential, willingness to use effective contraceptive method for the study duration and 6 months post-dosing.
* No surgery, radiotherapy or chemotherapy or any investigational agent within 30 days of study entry
* Signed written informed consent

Exclusion Criteria:

* Asecretory multiple myeloma
* Patients eligible and willing to undergo high dose chemotherapy followed by autologous stem cell transplantation
* Prior allogeneic transplantation
* Prior antibody or EGFR-pathway targeting therapy
* Severe cardiovascular disease like functionally restricting heart rhythm disturbance or heart malformation or severe hypertension, or cardiac insufficiency > NYHA-II
* HIV Infection, Hepatitis B or C
* Brain disorders, psychiatric illness
* Insufficient bone marrow reserve (Leucocytes < 1500/µl; Thrombocytes < 50000/µl)
* Creatinine-Clearance < 30 ml/min or Crea > 3.0 mg/dl
* Bilirubin > 2 mg/dl; ASAT, ALAT > 100 U/l
* Pregnancy (absence confirmed by serum/urine beta-HCG) or breast-feeding
* FEV1 < 50% of the reference value
* Active secondary malignancy
* Legal incapacity or limited legal capacity
* Having participated in another clinical trial or any investigational agent in the preceding 30 days
* Known allergic/hypersensitivity reaction to any compounds of the treatment
* Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Known drug abuse/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate (CR+PR+MR)at 16 weeks and during follow-up (every 3 months) | After 16 weeks

SECONDARY OUTCOMES:
Safety profile of Cetuximab +/- Dexamethasone | During 16 weeks of intervention and 8 weeks after
Freedom from treatment failure | From the date of registration until the first event or (if none occurs) until the date of the last determination of continuing complete/partial remission.
Progression-free survival | from the date of registration until first documentation of progression/relapse of disease or death related to MM
Overall survival | From the date of registration until the date of death from any cause or (if the patients is alive) until the date of last information.
Pharmacogenomic evaluation of response to treatment | After 16 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof. MD, Principal Investigator — University of Cologne
Locations (3):
- Germany (3):
  - University of Cologne, Department I of Internal Medicine, Cologne
  - Universtiy Hospital of Muenster, Internal Medicine A, Münster
  - University of Würzburg, Würzburg